CLINICAL TRIAL: NCT03090932
Title: Longitudinal Study of Innate Lymphoid Cells in Peripheral Blood in ALS
Status: Terminated | Type: Observational
Why Stopped: Study recruitment, data and sample collection terminated due to COVID-19. Data analysis continues.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Murdock, Research Investigator, University of Michigan
Other Study IDs: HUM00107546
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Innate lymphoid cells from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood draw — Research subjects will have two tubes of blood drawn, approximately 20mL.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a devastating neurodegenerative disorder characterized by progressive muscle weakness and eventual death. Studies demonstrate that the immune system plays a key role in ALS progression; however, the role of the immune system is unclear, as various aspects can play both a beneficial and detrimental role in the disease course. Attempts to universally suppress the immune system in ALS patients have at best had negligible effects on progression or at worst accelerated the disease. Thus, there is a critical need to identify immune cell populations to serve as biomarkers and therapeutic targets.

DETAILED DESCRIPTION:
Application - HUM00107546

Study Title:

Longitudinal Study of Innate Lymphoid Cells in Peripheral Blood in ALS

Full Study Title:

Longitudinal Study of Innate Lymphoid Cells in Peripheral Blood in ALS

If there are other U-M studies related to this project, enter the eResearch ID number (HUM#) or IRBMED Legacy study number. Examples of related projects include, but are not limited to:

00028826 - Epidemological Risk Factors and The Genetics of ALS

Principal Investigator:

* Benjamin Murdock, PhD

Study Team Members:

* Eva Feldman, MD, PhD Co-Investigator
* Stephen Goutman, MD Co-Investigator
* Claudia Figueroa-Romero, Research Investigator
* Crystal Pacut, Biorepository Coordinator
* Jayna Duell, Study Coordinator
* Blake Swihart, Study Coordinator
* Adam Patterson, Biostatistician

Project Summary:

Amyotrophic lateral sclerosis (ALS) is a devastating neurodegenerative disorder characterized by progressive muscle weakness and eventual death. Studies demonstrate that the immune system plays a key role in ALS progression; however, the role of the immune system is unclear, as various aspects can play both a beneficial and detrimental role in the disease course. Attempts to universally suppress the immune system in ALS patients have at best had negligible effects on progression or at worst accelerated the disease. Alternatively, augmenting or depleting specific immune cell populations in ALS mouse models alters the disease course and slows progression. Thus, there is a critical need to identify immune cell populations to serve as biomarkers and therapeutic targets.

Neuroinflammation is a hallmark of ALS in both human patients and mouse models. While clinical symptoms result from motor neuron degeneration, it is becoming increasingly clear that the immune system plays a key role in pathology. A variety of insults give rise to identical immune responses which go on to produce the characteristic clinical and histopathological manifestations of motor neuron disease. This makes the immune system an attractive target for therapeutics, as the wide variety of potential ALS sources all funnel through a common immunological pathway over the course of disease. The investigators recent studies have demonstrated that ALS patients have increased levels of several subpopulations of innate lymphoid cells (ILCs) in their peripheral blood. A subset of patients has ILC levels 5-10 times greater than those found in healthy control patients. The differences seen in the ILC levels in peripheral blood are much greater differences seen in other immune cell populations during ALS. Thus, these cell populations are attractive candidates for use as biomarkers or therapeutic targets.

The proposed study can be broken into three broad phases which will applicable to each patient: recruitment, sample collection, and analysis. Following diagnosis of disease, ALS patients who live within 1 hour of the University of Michigan will be called by our clinical coordinator and enrolled in the study (recruitment). Following enrollment in the study, each of the patients will be visited once every 28 ± 5 days for a year after the initial visit by a Michigan Institute for Clinical & Health Research (MICHR) clinical research unit; this unit will take 20 ml of blood per patient. Samples will then be returned to the University of Michigan. ILCs will be isolated from peripheral blood using fluorescence-activated cell sorting (FACS) and the mRNA of each ILC population will be collected and cytokine production analyzed using multiplex (analysis). On the day of collection, a clinician or clinical coordinator from the University of Michigan Comprehensive ALS Clinic (UMCAC) will contact the patient to complete an ALSFRS-R questionnaire to assess the physical deterioration of the patients.

The study will also incorporate control subjects. The control subjects will have blood taken once a month for 12 total visits over 36 months, but will not complete the ALSFRS-R questionnaire as they will not have been diagnosed with ALS and therefore the questionnaire does not fit; 20ml of blood will be taken per visit.

Subjects need to live within approximately 60 miles of the University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Clinically definite, probable, probable laboratory supported, or possible ALS by El Escorial criteria
* Fluency in English at the 6th grade level or higher.
* Able to communicate sufficiently well by speaking
* Able to communicate over the phone.
* Capable of providing informed consent.
* Lives geographically accessible to the University of Michigan

Exclusion Criteria:

* Unable to provide informed consent.
* Clinically significant dementia, as judged by the site investigator.
* Other neurological or psychiatric disorders which are expected to impair cognitive function.
* Other serious and uncontrolled medical disorders.
* History of autoimmune disease.
* Use of prednisone, IVIG, or immunosuppression within the last 12 months.
* Not geographically accessible to the University of Michigan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS patients (200) and matched controls (75)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Total number of classical NK (natural killer) cells; total number of CD3+ CD4+ CD8+ cells | Every 28 days (+/- 5 days) for 12 total visits over 36 months
  Total number of classical NK cells; total number of CD3+ CD4+ CD8+ cells

SECONDARY OUTCOMES:
Cytokine expression | Every 28 days (+/- 5 days) for 12 total visits over 36 months
  Cytokine expression levels of these cell populations using qPCR, RNA-Seq, or Luminex.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Murdock, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided